CLINICAL TRIAL: NCT01111825
Title: A Phase I/II Trial of Temsirolimus Plus Neratinib for Patients With Metastatic HER2-Amplified or Triple Negative Breast Cancer
Brief Title: Temsirolimus Plus Neratinib for Patients With Metastatic HER2-Amplified or Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-005
Record Dates: First submitted 2010-04-22; First posted 2010-04-28 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: HKI-272 (NERATINIB); TEMSIROLIMUS (CCI-779); HER2-Amplified; Triple-negative; invasive adenocarcinoma; 10-005; Nerlynx; PB-272
MeSH Terms: conditions — Breast Neoplasms | interventions — temsirolimus; neratinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Temsirolimus plus Neratinib (Experimental): This is an open-label, single arm, dose-escalation phase I-II study to determine the maximum tolerated dose (MTD) of temsirolimus with daily neratinib, and to determine the safety and efficacy of this combination when given to patients with advanced breast carcinoma. Patients with trastuzumab-refractory HER2-amplified disease or triple negative disease will be enrolled in both phases of this clinical trial.
  Interventions: Drug: Temsirolimus; Drug: Neratinib

INTERVENTIONS:
Drug: Temsirolimus — 28 day treatment cycle Phase 1
  * Weekly intravenously (IV) on days 1, 8, 15, and 22
  * Starting dose 8 mg IV weekly (dose level 1). Three patients initially enrolled in each cohort
  Phase 2
  * Dose escalation cohort - 8 mg IV weekly on Days 1, 8, 15, and 22, and then 15 mg IV weekly starting on Day 29
  * HER2-amplified and Triple negative - 8 mg IV weekly on Days 1, 8, 15, and 22
  Other Names: Torisel
Drug: Neratinib — 28 day treatment cycle
  • 240 mg orally daily
  Other Names: Nerlynx

SUMMARY:
This is an open-label, single arm, multi-center, multi-national, adaptive design, dose-escalation Phase 1/2 study to determine the maximum tolerated dose (MTD) of temsirolimus with daily neratinib, and to determine the safety and efficacy of this combination when given to patients with advanced breast carcinoma, specifically trastuzumab-refractory HER2-amplified disease or triple-negative disease.

DETAILED DESCRIPTION:
Phase I Design A standard, 3+3, dose escalation schedule to determine the MTD of temsirolimus in combination with neratinib with no intrapatient dose escalation and a starting dose of temsirolimus 8 mg administered intravenously (IV) weekly (dose level 1) and three patients enrolled in each cohort.

Phase II Design The phase II portion of this trial is comprised of three cohorts. Two of the cohorts utilized a Simon two-stage design to determine the sample size to assess the efficacy of temsirolimus when administered in combination with neratinib: HER2-amplified and triple negative breast cancer. The third cohort was a single stage design with HER2-amplified patients and dose escalation.

ELIGIBILITY:
Inclusion Criteria:

Phase I HER2-amplified Cohort

* HER2 overexpression and/or amplification as determined by immunohistochemistry (3+) or fluorescence in situ hybridisation (FISH) (≥2.0)
* Previously received trastuzumab as part of a regimen in the adjuvant or metastatic setting with evidence of progression. Washout period for trastuzumab of 14 days.
* May have previously received lapatinib as part of a regimen in the adjuvant or metastatic setting with evidence of progression of disease. Washout period for lapatinib of 14 days.
* Radiographic progression of disease while on treatment with trastuzumab or lapatinib as defined by RECIST 1.1 criteria.
* No restriction on prior chemotherapy regimens for advanced stage disease. No restriction for prior hormonal therapy. No concurrent use of endocrine therapy is permitted.

Phase II HER2-amplified Cohort

* HER2 overexpression and/or amplification as determined by immunohistochemistry (3+) or FISH (≥2.0).
* Previously received trastuzumab as part of a regimen in the adjuvant or metastatic setting with evidence of progression. Washout period for trastuzumab of 14 days.
* May have previously received lapatinib as part of a regimen in the adjuvant or metastatic setting with evidence of progression of disease. Washout period for lapatinib of 14 days.
* Radiographic progression of disease while on treatment with trastuzumab as defined by RECIST 1.1 criteria.
* Prior therapy inclusion: no more than four prior chemotherapy regimens allowed for advanced stage disease. No restriction for prior hormonal therapy. No concurrent use of endocrine therapy is permitted.

Phase II Triple-negative Cohort - As of 2/10/12, this cohort is closed to accrual

* Invasive adenocarcinoma negative for estrogen receptor (<5%) and progesterone receptor (<5%) expression and a lack of HER2 overexpression and/or amplification as determined by immunohistochemistry (<3+) or FISH (<2.0).
* Prior therapy inclusion: no more than four prior chemotherapy regimens allowed for advanced stage disease. No restriction for prior hormonal therapy. No concurrent use of endocrine therapy is permitted.

Phase II HER2-Positive Cohort with dose escalation

* HER2 overexpression and/or amplification as determined by immunohistochemistry (IHC) (3+) or FISH (≥2.0).
* Previously received trastuzumab as part of a regimen in the adjuvant or metastatic setting with evidence of progression. Washout period for trastuzumab of 14 days.
* May have previously received lapatinib as part of a regimen in the adjuvant or metastatic setting with evidence of progression of disease. Washout period for lapatinib of 14 days.
* Radiographic progression of disease while on treatment with trastuzumab as defined by RECIST v 1.1.
* Prior therapy inclusion: no restriction on prior chemotherapy regimens for advanced stage disease. No restriction for prior hormonal therapy. No concurrent use of endocrine therapy is permitted.

Inclusion Criteria for all subjects (HER2-Amplified and Triple-negative)

* Patients with a diagnosis of invasive adenocarcinoma of the breast confirmed by histology or cytology at MSKCC.
* Metastatic disease that is or has been pathologically documented.
* At least one measurable metastatic lesion according to RECIST 1.1 criteria. Ascites, pleural effusions, and bone metastases are not considered measurable. Minimum indicator lesion size ≥ 10 mm by helical CT or ≥ 20 mm by conventional techniques.
* Pathological nodes must be ≥ 15 mm by the short axis to be considered measurable.
* Age ≥ 18, as no dosing or adverse event data are currently available on the use of neratinib or temsirolimus in patients <18 years of age, children are excluded from this study.
* Patients must be willing to discontinue sex hormonal therapy, e.g., birth control pills, hormonal replacement therapy, prior to enrollment. Women of childbearing potential must consent to effective contraception while on treatment and for a period thereafter.
* Negative serum human chorionic gonadotropin pregnancy test for premenopausal women of reproductive capacity and for women less than 12 months after menopause.
* Asymptomatic, central nervous system metastases are permitted if patients remain clinically stable after discontinuation of steroids and anticonvulsants for 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
* Patients must have normal organ and marrow function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5x institutional upper limit of normal except for patients with liver metastases. For patients with liver metastases, AST/ALT/Alkaline phosphatase ≤5.0x institutional upper limit of normal. Total bilirubin within institutional limits except for patients with liver metastases. For patients with liver metastases, total bilirubin ≤1.5x institutional upper limit of normal. Creatinine clearance within normal limits or ≥ 60 mL/min, prothrombin time and partial thromboplastin time ≤1.5x institutional upper limit of normal except for patients on Coumadin or low molecular weight heparin, leukocytes ≥3,000/μl, absolute neutrophil count ≥1,000/μl, and platelets ≥75,000/μl
* Able to swallow and retain oral medication.

The following criteria were removed for all patients in Protocol Amendment 10, and are only applicable to first 34 HER2+ patients in Phase 2 who are not subject to dose-escalation of temsirolimus:

* Able and willing to consent for biopsy of metastatic breast cancer prior to treatment. Consent to preservation of frozen and fixed samples of tumor cores for evaluation. (HER2-amplified patients who have previously provided samples of metastatic breast cancer as part of institutional review board #06-163 will be exempt)
* Consent to evaluation of primary tumor biopsy specimen.

Exclusion Criteria:

* Potential subjects will be excluded from enrollment into this study if they meet any of the following criteria:
* Patients receiving any concurrent anticancer therapy or investigational agents with the intention of treating breast cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to neratinib or temsirolimus.
* Unable to consent to biopsy of metastatic disease or for whom a biopsy would be medically unsafe.
* Women who are pregnant or breast feeding.
* Life expectancy <3 months.
* Completion of previous chemotherapy regimen <3 weeks prior to the start of study treatment. Prior hormonal therapy must be discontinued prior to treatment start. Biologic therapy with bevacizumab for the treatment of metastatic disease must be discontinued ≥3 weeks from the start of protocol treatment.
* Concurrent radiotherapy is not permitted for disease progression on treatment on protocol, but might be allowed for pre-existing non-target lesions with approval from the principal investigator of the trial.
* Concurrent medical conditions which may increase the risk of toxicity, including ongoing or active infection, history of significant bleeding disorder unrelated to cancer (congenital bleeding disorders, acquired bleeding disorders within one year), HIV-positive or active hepatitis.
* History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, and left ventricular ejection fraction less than 50% measured by a multigated blood pool imaging of the heart (MUGA scan) or an echocardiogram (ECHO).
* QT corrected interval > 0.47 seconds.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease.
* History of an invasive second primary malignancy diagnosed within the previous 3 years, except for stage I endometrial or cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures are necessary to participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma Biotechnology, Study Director — Puma
Locations (12):
- United States (4):
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Weill Cornell Medical College - New York - Presbyterian Hospital, New York, New York
- Roskilde Hospital, Roskilde, Denmark
- Institut Gustave Roussy, Villejuif, France
- UNIMED Medical Institute, Wan Chai, Hong Kong
- Spain (3):
  - Hospital Universitario Sant Joan de Reus, Tarragona, Reus
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
- United Kingdom (2):
  - Edinburgh Cancer Center, Western General Hospital, Edinburgh
  - The Royal Marsden NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Phase I, HER - Amplified (HER2-Positive) cohort
- Phase 2 Triple -ve: Phase 2, Triple - Negative cohort
- Phase 2 HER2+: Phase 2, HER2 - Amplified (HER2-Positive) cohort
- Phase 2 HER2+ Dose Esc: Phase 2, HER2 - Positive cohort with dose escalation
Period: Overall Study
Arm/Group | Phase 1 | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Started | 8 | 6 | 37 | 48
Completed (Completed means completed study or died.) | 5 | 5 | 29 | 27
Not Completed | 3 | 1 | 8 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Adverse Event | 2 | 1 | 4 | 0
Not completed — Disease Progression | 1 | 0 | 0 | 0
Not completed — Discontinuation by Sponsor | 0 | 0 | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc | Total
Number analyzed (Participants) | 8 | 6 | 37 | 48 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 34 | 39 | 85
  >=65 years | 1 | 1 | 3 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (10.4) | 53.5 (13.0) | 52.0 (8.3) | 53.2 (11.0) | 52.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 37 | 47 | 98
  Male | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) (Phase II)
Description: ORR is defined as proportion of subjects who achieved confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  A complete or partial response must be confirmed no less than 4-weeks after the criteria for response are initially met.
Time Frame: From enrollment date to first documented response, or last tumor assessment, assessed up to two years
Population: Intent to Treat (ITT) population (all enrolled subjects) for the Phase II portion of the study. Per protocol, Phase I data was not included in efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Number analyzed (Participants) | 6 | 37 | 48
Participants | 0 | 5 | 14

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Defined as the proportion of patients who achieved objective response (CR or PR) or SD for at least 24 weeks per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
  Clinical Benefit (CB) = CR + PR + SD >= 24 weeks.
Time Frame: From enrollment date to first documented response, or last tumor assessment, assessed up to two years
Population: ITT population (all enrolled subjects) for the Phase II portion of the study. Per protocol, Phase I data was not included in efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Number analyzed (Participants) | 6 | 37 | 48
Participants | 0 | 8 | 19

3. Secondary Outcome: Duration of Response (DOR)
Description: Measured from the time at which measurement criteria were first met for CR or PR (whichever status was recorded first), until the date of first recurrence, Progressive Disease (PD), or death was objectively documented, taking as a reference for PD the smallest measurements recorded since enrollment, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progressive Disease (PD), At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, and/or the appearance of one or more new lesions.
Time Frame: From first response to first PD or death, assessed up to two years.
Population: Patients who were enrolled and responded in the Phase II portion of the study. Per protocol, Phase I data was not included in efficacy analysis.
  Note, no subject in Phase II triple negative cohort had a response. Therefore, no participants were analyzed for DOR.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Number analyzed (Participants) | 0 | 5 | 14
Participants
  0 to <3 months | 0 | 1 | 2
  3 to <6 months | 0 | 2 | 1
  6 to <9 months | 0 | 0 | 6
  9 to <12 months | 0 | 2 | 2
  12+ months | 0 | 0 | 3

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as time from date of enrollment until the first disease recurrence or progression or death due to any cause; censored at the last assessable evaluation or at the initiation of new anti-cancer therapy. Disease assessment is based on investigator tumor assessments. If no post-baseline tumor assessment then censored at enrollment date.
Time Frame: From date of enrollment until the date of first documented progression, or date of death from any cause, whichever came first, assessed up to two years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Number analyzed (Participants) | 6 | 37 | 48
months | 1.8 [1.8 to 2.0] | 4.8 [2.7 to 8.4] | 6.0 [3.7 to 8.3]

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from enrollment to death due to any cause; censored at the date last known alive.
Time Frame: From enrollment to date of death from any cause, or end of long term follow-up, assessed up to three years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 HER2+ Dose Esc
Number analyzed (Participants) | 48
months | 17.8 [13.4 to NA] — Upper limit of confidence interval is not estimable.

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, assessed up to two years.
Description: Safety Population
Arm/Group | Phase 1 | Phase 2 Triple -ve | Phase 2 HER2+ | Phase 2 HER2+ Dose Esc
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/6 | 12/37 | 20/48
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 37/37 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=8) | Phase 2 Triple -ve (N=6) | Phase 2 HER2+ (N=37) | Phase 2 HER2+ Dose Esc (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Cerebral disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=8) | Phase 2 Triple -ve (N=6) | Phase 2 HER2+ (N=37) | Phase 2 HER2+ Dose Esc (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 3 | 2
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 8
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 2 | 7 | 21
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 35 | 40
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Nausea (Gastrointestinal disorders) | 6 | 5 | 18 | 20
Stomatitis (Gastrointestinal disorders) | 5 | 4 | 25 | 29
Vomiting (Gastrointestinal disorders) | 3 | 3 | 9 | 23
Asthenia (General disorders) | 0 | 0 | 0 | 18
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 1
Fatigue (General disorders) | 6 | 3 | 20 | 9
Oedema peripheral (General disorders) | 2 | 1 | 2 | 9
Pain (General disorders) | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 6 | 4
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 3
Localised infection (Infections and infestations) | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 5
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 4 | 4
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Stoma site ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 4
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 3
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 4
Weight decreased (Investigations) | 3 | 2 | 5 | 6
Weight increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 6 | 19
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 6
Dizziness (Nervous system disorders) | 1 | 0 | 6 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 4 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 11
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 7 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 4
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 10
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 7 | 4
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 17 | 21
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 2 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 1 | 2
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less